CLINICAL TRIAL: NCT05958797
Title: Efficacy and Safety of Chloroquine for Plasmodium Vivax in the Philippines in 2016.
Brief Title: TES of Chloroquine for Pv in the Philippines in 2016
Acronym: TES
Status: Completed | Type: Observational
Sponsor: Research Institute for Tropical Medicine, Philippines (Other Government)
Collaborators: World Health Organization (Other)
Responsible Party: Principal Investigator, Fe Espino, Principal Investigator, Head of Parasitology Department, Research Institute for Tropical Medicine, Philippines
Other Study IDs: 2003-25-12_2016
Record Dates: First submitted 2023-06-30; First posted 2023-07-25 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Malaria; Vivax Malaria; Recrudescence
Keywords: malaria; TES; Plasmodium vivax; Chloroquine
MeSH Terms: conditions — Malaria; Malaria, Vivax; Recurrence | interventions — Chloroquine; Primaquine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Capillary blood (malaria blood film and filter paper)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Patients detected with Plasmodium vivax (Chloroquine): Patients with mono-infection of Plasmodium falciparum with ≥ 250 per µl
  Interventions: Drug: Chloroquine; Drug: Primaquine

INTERVENTIONS:
Drug: Chloroquine — Chloroquine will be administered according to body weight at a total dose of 25 mg base/kg over 3 days (10 mg base/kg on Day 0; 10 mg base/kg on Day 1 and 5 mg base/kg on Day 2). Correct drug dosage will be determined using the dosing chart (in accordance
Drug: Primaquine — For Pf patients, primaquine at 0.75 mg base/kg body weight single dose will be given on Day 3 for Pf patients; For Pv patients primaquine will be withheld for 28 days and will be given after Day 28 follow-up, at 0.25 mg base/kg per day for 14 days.

SUMMARY:
Chloroquine (CQ) is officially used as a first-line drug of Plasmodium vivax malaria in the Philippines. In this study, the therapeutic efficacy of CQ for the treatment of uncomplicated P. vivax malaria in three (3) municipalities (Bataraza, Brooke's Point and Rizal) of Palawan was evaluated using the World Health Organization protocol with a follow-up of 28 days and additional 2 days (Day 31 and 34) for hemoglobin monitoring after primaquine treatment. Study subjects were febrile individuals between > 6 months old and 59 years old with confirmed uncomplicated P. vivax infections. Chloroquine was administered according to body weight at a total dose of 25 mg/kg over 3 days (10 mg/kg on Day 0; 10 mg/kg on Day 1 and 5 mg/kg on Day 2), and primaquine following the National Treatment Guidelines. During the 1 year period that this report covers, there were 8,305 individuals were screened.

DETAILED DESCRIPTION:
In 2002, the Philippines changed its antimalarial drug policy to a combination treatment, CQ+SP as the 1st-line treatment and artemether-lumefantrine as the 2nd-line treatment. The DOH prescribed the use of an artemether-lumefantrine (AL) combination as the second-line drug, limiting its use only in the treatment of confirmed Plasmodium falciparum, until a further study on its efficacy was done before making it the first-line treatment. Consequently, AL became the first-line drug for falciparum malaria in the 2009 revised drug policy. The DOH in the past 6 years (2002-2007) adopted the use of AL in the highly endemic areas of the country and conducted therapeutic efficacy studies (TES) in 3 sentinel sites: Kalinga-Isabela, Palawan and several Mindanao provinces, showing 97-100% efficacy. Whereas CQ+SP showed variability and declining efficacy, results ranged from 70%-95% (CARAGA region). In Sultan Kudarat province, results in 2006-2007 showed 90% efficacy of CQ+SP and 96% for AL for falciparum malaria.

In the 2009 drug policy, chloroquine (CQ) remains the primary treatment for P. vivax malaria, with primaquine as an anti-relapse drug. Previous studies (1999-2005) elsewhere in the country have shown 100% efficacy of CQ or the CQ+PQ combination. Furthermore, in the 2013-2014 study, recurrence of parasitemia was observed in two of 75 enrolled patients in Palawan. This study updates the drug efficacy for P. vivax malaria in the country.

STUDY OBJECTIVES The general objective of this study is to assess the therapeutic efficacy and safety of chloroquine for the treatment of P. vivax infections in Palawan province, the Philippines in 2016.

The specific objectives are:

1. To measure the clinical and parasitological efficacy of Chloroquine among patients aged between > 6 months and 59 years old suffering from vivax malaria, by determining the proportion of patients with Early Treatment Failure (ETF), Late Clinical Failure (LTF), Late Parasitological Failure (LPF), or with an Adequate Clinical and Parasitological Response (ACPR) as indicators of efficacy;
2. To evaluate the incidence of adverse events;
3. To formulate recommendations to enable the Department of Health to make informed decisions about the possible need for updating of the current national antimalarial treatment guidelines.

MATERIALS AND METHODS. The design of this surveillance study is a one-arm, prospective evaluation of the clinical and parasitological response to directly observed treatment for vivax malaria. Individuals with vivax malaria who met the study inclusion criteria were enrolled, treated on-site with CQ+PQ, and monitored for a period of 28 days. The follow-up consisted of a fixed schedule of check-up visits and corresponding clinical and laboratory examinations. Study patients had been classified as therapeutic failures (early or late) or adequate responders based on the results of these assessments. The proportion of patients experiencing a therapeutic failure during the follow-up period had been used to estimate the efficacy of the study drug(s). Polymerase Chain Reaction (PCR) analysis will also help distinguishes between a true recrudescence due to treatment failure and episodes of re-infection.

Barangay Health Workers and Barangay Malaria Microscopists were mobilized to recruit febrile patients (patients with body temperature ≥37.5 °C). Screened individuals were re-examined at the main health center for malaria symptoms, body temperature, and weight. All laboratory procedures and tests were carried out by trained staff.

STUDY AREA / SETTINGS. The study was conducted in the Rural Health Units (RHU) of Rizal, Bataraza, and Brookes Point. Several factors influenced the selection of sites: (a) adequate numbers of patients with symptomatic, P. vivax; (b) willingness and availability of the selected healthcare facility staff to participate in the trial and to support the work with laboratory space; (c) access of patients to the health facility for weekly follow-ups; and (d) willingness of the Municipality Health Officer (MHO), the nurse and a trained Medical Technologist to take responsibility for conducting the trial, and security.

STUDY PARTICIPANTS. The population of interest consisted of patients aged between > 6 months to 59 years old diagnosed with uncomplicated vivax malaria attending the study health clinic and having given, or whose parents or legal guardians have given informed consent for study inclusion and assent in children as appropriate.

SAMPLE SIZE. Treatment failure to CQ in the area being 0-5%, 5% has been chosen as the estimated therapeutic failure rate of the drug. At a confidence level of 95% and with precision around the estimate of 10%, 18 patients will be needed. With a 20% increase to allow losses to follow-up and withdrawals during the 28-day follow-up period, 22 patients need to be included. But in order for the sample to be representative, a minimum of 50 P. vivax patients need to be included and a maximum of 75 Plasmodium vivax were enrolled.

SAMPLING TECHNIQUE. All individuals who consulted at the selected rural health units met the inclusion criteria and had none of the exclusion criteria included in the study.

DATA MANAGEMENT. The principal investigator has ensured that the study protocol is strictly adhered to throughout and that all data are collected and recorded correctly on the CRF. Laboratory and clinical data have been recorded on a daily basis in the CRF designed for the study. Data that are derived from source documents are consistent with the source documents or the discrepancies were explained. Any changes or corrections to a CRF were dated and explained and did not obscure the original entry. All CRF was checked for completeness. After the study was completed, data were entered into a database using double independent data entry. The data were stored in a computer database maintaining confidentiality in accordance with the national data legislation.

ETHICAL CONSIDERATIONS. Participants were recruited after the study received favorable approval of the protocol, participant information sheet, and written informed consent form from RITM Institutional Review Board (IRB). The study document versions given written approval by the IRB were used. The study was carried out according to the ethical guidelines in the Declaration of Helsinki (version 2008), applicable guidelines of ICH-GCP (E6); and applicable regulations of the Department of Health, Manila. The participant's written informed consent was secured before enrolment and prior to initiating procedures specific to this study. For potential participants below 18 years old, this consent was obtained from the either parent or a legally accepted guardian. An independent witness was present during the process of obtaining informed consent from a participant or parents/legal guardian who was illiterate.

ELIGIBILITY:
Inclusion Criteria:

* Above 6 months old to 59 years old;
* Mono-infection with P. vivax (≥250/ul)
* Axillary temperature ≥37.5 °C or oral/rectal temperature of ≥38 °C;
* Glucose-6-dehydrogenase (G6PD) test normal for vivax patients if available
* Ability to swallow medication;
* Ability and willingness to comply with the study protocol for the duration of the study and to comply with the study visit schedule;
* Informed consent from the patient or from a parent or legal guardian in the case of children less than 18 years old;
* Informed assent from any minor participant aged 12 - 17 years; and
* Consent for pregnancy testing from females of child-bearing potential and from their parent or guardian if under 18 years old.

Exclusion Criteria:

* Presence of general danger signs among children <5 years old or other signs of severe and complicated falciparum malaria according to current WHO definitions
* Mixed Plasmodium species;
* Presence of severe malnutrition
* Presence of febrile conditions due to diseases other than malaria (measles, acute lower tract respiratory infection, severe diarrhea with dehydration, etc.), or other known underlying chronic or severe diseases (e.g. cardiac, renal, hepatic diseases, HIV/AIDS)
* History of hypersensitivity reactions to any of the drug(s) being tested or used as alternative treatment.

Ages: 6 Months to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The population of interest consists of patients aged between > 6 months to 59 years old diagnosed with uncomplicated vivax malaria attending the study health clinic, and having given, or whose parents or legal guardians have given informed consent for study inclusion and assent in children as appropriate.
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2016-01-04 (Actual); Primary Completion 2016-12-29 (Actual); Study Completion 2016-12-29 (Actual)

PRIMARY OUTCOMES:
Number of Patients with Early Treatment Failure (ETF) | Day 1-3
  The number of patients with the following criteria based on microscopy results without PCR:
  * Development of danger signs or severe malaria on day 1, day 2, or day 3 in the presence of parasitemia;
  * Parasitaemia on day 2 higher than day 0 count irrespective of axillary temperature;
  * Parasitaemia on day 3 with axillary temperature ≥37.5 ºC;
  * Parasitaemia on day 3 ≥25% of count on day 0.
Number of Patients with Late Clinical Failure (LCF) | Day 4-28
  The number of patients with the following criteria based on microscopy results without PCR:
  * Development of danger signs or severe malaria on day 1, day 2, or day 3 in the presence of parasitemia;
  * Parasitaemia on day 2 higher than day 0 count irrespective of axillary temperature;
  * Parasitaemia on day 3 with axillary temperature ≥37.5 ºC;
  * Parasitaemia on day 3 ≥25% of count on day 0.
Number of Patients with Late Parasitological Failure (LPF) | Day 7-28
  The number of patients with the presence of parasitemia on any day from day 7 to day 28 and axillary temperature <37.5 ºC, without previously meeting any of the criteria of Early Treatment Failure or Late Clinical Failure.
Number of Patients with Adequate Clinical and Parasitological Response (ACPR) | Day 0-28
  The number of patients with absence of parasitemia on day 28 irrespective of axillary temperature without previously meeting any of the criteria of Early Treatment Failure or Late Clinical Failure or Late Parasitological Failure.

CONTACTS AND LOCATIONS:
Overall Officials: Fe Esperanza Caridad J Espino, MD, PhD, Principal Investigator — Research Institute for Tropical Medicine

IPD SHARING:
Plan to Share IPD: Yes
The IPD will be shared with Data Transfer Agreement and IRB Approval
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data information will be provided upon request
Access Criteria: Data Transfer

REFERENCES:
- [Background] Council for International Organizations of Medical Sciences. International ethical guidelines for biomedical research involving human subjects. Bull Med Ethics. 2002 Oct;(182):17-23. PMID 14983848
- [Background] World Medical Association. World Medical Association Declaration of Helsinki: ethical principles for medical research involving human subjects. JAMA. 2013 Nov 27;310(20):2191-4. doi: 10.1001/jama.2013.281053. No abstract available. PMID 24141714

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-19): https://cdn.clinicaltrials.gov/large-docs/97/NCT05958797/Prot_SAP_000.pdf